CLINICAL TRIAL: NCT05196243
Title: A New Multimodal Imaging Technique Based on Pathological and Genomic Characteristics of Gastrointestinal Mucosa
Brief Title: Multimodal Imaging Based on Pathological and Genomic Characteristics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: Multi-imaging
Record Dates: First submitted 2022-01-05; First posted 2022-01-19 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Mitochondrial DNA Mutation; Endoscopy
Keywords: Mitochondrial DNA Mutation; Single cell sequencing; Molecular pathology; multimodal imaging; holography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Mucosal tissues or cells of gastritis, gastric cancer, intestinal polyps and colorectal cancer obtained by endoscopic biopsy or resection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: Study on the genomic and molecular pathological characteristics of gastrointestinal mucosal lesions
  Interventions: Other: Patients diagnosed as gastrointestinal mucosal lesions
- Control Group: Study on the genomic and molecular pathological characteristics of normal gastrointestinal mucosa

INTERVENTIONS:
Other: Patients diagnosed as gastrointestinal mucosal lesions — Patients diagnosed as gastritis, gastric cancer, intestinal polyps and colorectal cancer
  Groups: Study Group

SUMMARY:
Mitochondrial DNA mutations in normal gastric tissue, early gastric cancer and advanced gastric cancer were identified by single cell sequencing, and the origin of gastric stem cells was traced and new molecular markers were found. At the same time, organize industry-university-research-medical inspection joint research, aiming at the advanced layout of new structural and functional imaging technologies, combined with some new imaging technologies, such as holography, fluorescence, etc., to explore and develop a new composite endoscopic imaging technology that is advanced, original and suitable for China's national conditions, in order to develop a prototype of multimodal structural and functional imaging digestive endoscope without contrast agent.

DETAILED DESCRIPTION:
In this study, on the basis of previous work, aiming at the visualization of key molecular functions of gastric cancer, a full-chain digestive endoscopic diagnosis system was constructed by using cross-scale medical imaging technology. Mitochondrial DNA mutations in normal gastric tissue, early gastric cancer and advanced gastric cancer were identified by single cell sequencing, and the origin of gastric stem cells was traced and new molecular markers were found. The tissue characteristics are analyzed by the full spectrum imaging device, and the location, distribution and aggregation of key molecules on the cell membrane are observed by the high resolution imaging device, so as to develop an imaging probe with high labeling efficiency and biosafety, and to explore its clinical application to realize the information fusion of structural and functional imaging in the evolution and diagnosis and treatment of gastrointestinal tumors. The structural heterogeneity and molecular heterogeneity of gastrointestinal tumors are clarified from the macro-micro levels, and the full-scale imaging system with the most comprehensive visualization and resolution ability is established from multi-information dimensions and multi-imaging scales.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis or suspected diagnosis of one of the following common digestive mucosal diseases: gastritis, gastric cancer, colorectal polyps, bowel cancer
2. Written informed consent

Exclusion Criteria:

1. Patients with cardiovascular and cerebrovascular diseases, or patients with severe impairment of liver, kidney and hematopoietic system
2. Mental patients
3. Hemorrhagic diseases
4. Platelet count < 50 × 10 ^ 9 / L
5. Allergic constitution
6. unable to tolerate or cooperate with endoscopy
7. Patients with serious complications, such as intestinal obstruction, intestinal perforation, toxic colonic dilatation, colorectal cancer, etc.
8. Pregnant or lactating women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People diagnosed or suspected of one of the following common digestive mucosal diseases: gastritis, gastric cancer, colorectal polyps, colorectal cancer
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Single cell sequencing and identification of mitochondrial DNA variation in gastrointestinal lesions | 1 month
  Single cell sequencing and identification of mitochondrial DNA mutations in gastrointestinal lesions were carried out to trace the clonal origin of cells and look for molecular markers
To explore the multimodal imaging technique for the diagnosis of gastrointestinal mucosal lesions | 1 month
  The tissue characteristics are analyzed by the full spectrum imaging device, the location, distribution and aggregation of key molecules on the cell membrane are observed by the high resolution imaging device, the imaging probe with high labeling efficiency and biosafety is developed, and the clinical application is discussed. in order to realize the information fusion of structural and functional imaging in the process of gastrointestinal tumor evolution and diagnosis and treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Liu, MD, Principal Investigator — Beijing 302 Hospital
Locations (1):
- The First Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality, China